CLINICAL TRIAL: NCT03673553
Title: The Unite Care of Fibromyalgia. The Experience of the Patients and the Professionals.
Brief Title: The Multidisciplinary Treatment of Fibromyalgia.
Status: Completed | Type: Observational
Sponsor: Institut Investigacio Sanitaria Pere Virgili (Other)
Responsible Party: Principal Investigator, Verge Cinta_Carlos Lopez, Principal Investigator, Institut Investigacio Sanitaria Pere Virgili
Other Study IDs: CEIC-1488
Record Dates: First submitted 2018-09-06; First posted 2018-09-17 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Fibromyalgia; Pain; Treatment; Quality of Life
Keywords: fibromyalgia; pain; quality of life; multidomal treatment
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Association of people with fibromyalgia: Control group included people affiliated to the FM Patient Association of Terres de l'Ebre, Spain.
  Interventions: Other: Association of people with fibromyalgia
- Multimodal treatment of patients with FM: The intervention group was made up of patients from the specialist FM Unit in the Hospital of Lleida, Spain.
  Interventions: Other: Multimodal treatment of patients with FM

INTERVENTIONS:
Other: Multimodal treatment of patients with FM — The intervention group took part in 2.5-hour sessions of MRT once a week for 10 weeks. This intervention combined physical exercise with stretching. Health education was geared towards pain management, the pathology itself, healthy habits, insomnia, postural correction and ergonomics. The psychological approaches used in the MRT were problem-solving therapy, cognitive behavioural therapy and sophrology. Given the diversity of the sessions, they were directed by a rheumatologist, a nurse, a psychologist, and a physiotherapist. If the patient needed their pharmacological treatment to be altered, they were offered an appointment with the rheumatologist.
  Groups: Multimodal treatment of patients with FM
Other: Association of people with fibromyalgia — The control group attended the activities organised by the association of people with FMS. These consisted of a weekly 1-hour session of group psychology and a weekly 2-hour session of handicrafts for 10 weeks.
  Groups: Association of people with fibromyalgia

SUMMARY:
Background Fibromyalgia is a pathology characterised by chronic pain that harms people's quality of life. This pathology requires an MRT that combines pharmacological and non-pharmacological treatments. Currently, FPAs are important to society not only by offering activities that improve fibromyalgia symptomatology but also by increasing public awareness of the disease. The present study compares the effectiveness of a multimodal rehabilitation treatment (MRT) with that of the activities of a fibromyalgia patient association (FPA), and identifies the patient characteristics that can interfere with the success of interventions.

Methods The quasi-experimental study selected forty-six older adults with fibromyalgia. The intervention group (n = 23) received pharmacological treatment, physical exercise, education, psychological therapies and Caycedian sophrology, while the control group (n = 23) carried out group psychological sessions and handicraft-based activities. Data collection included sociodemographic measures and responses to the Fibromyalgia Impact Questionnaire (FIQ). Participants were assessed pre- and post-intervention.

DETAILED DESCRIPTION:
A descriptive analysis of the sociodemographic characteristics of the intervention and control groups was done. Qualitative variables were expressed as percentages, and quantitative variables were summarised as the median and interquartile range.

Shapiro-Wilk tests indicated that the dependent variables were not normally distributed (p < .05), so non-parametric statistical analyses were subsequently performed. The difference between the medians of the two patient groups was examined with the Mann-Whitney U test. Qualitative variables were compared with the chi-squared or Fisher's exact test, as appropriate.

Being a quasi-experimental study, without randomization of patients, the existence of initial pre-intervention differences in the dimensions evaluated by the FIQ scale between the two patient groups was tested with the Mann-Whitney U test. For the dimensions that showed significant pre-intervention group differences, the medians of the post- and pre-intervention differences between the two patient groups were tested. For those dimensions of the FIQ that showed no pre-intervention differences, the post-intervention values were compared. The changes in the FIQ score and its dimensions before and after the intervention in both groups were assessed using the Wilcoxon test.

Additionally, we carried out univariate and multivariate logistic regression analyses to identify the relationships between the independent variables studied and the improvement variable (increase, or not, of at least 8.1 points in the FIQ score after the intervention).

Finally, the sample was stratified by educational level (primary versus secondary/university studies) and age (younger than 60 years or 60+ years). The pre- and post-intervention scores were compared using the Mann-Whitney U test and the differences in each group were analysed with the Wilcoxon test.

ELIGIBILITY:
Eligibility Criteria inclusion intervention group:

* to be diagnosed with FM
* to be between 18 and 80 years old
* be a patient of the unit care of FM
* the patients have to participate in nine of the treatment sessions
* the patients have to make the first visit in the unit care of FM during 2016

Eligibility Criteria inclusion control group:

* to be diagnosed with FM
* to be between 18 and 80 years old
* to be a member of the FM Patient Association of Terres de l'Ebre

Eligibility Criteria exclusion control intervention and group:

* not understanding Catalan or Spanish
* not providing correct contact data

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample size was calculated on the basis of accepting an alpha risk of less than 0.05 and a beta risk of less than 0.20. The calculation indicated that 23 subjects each in the intervention and control groups were needed to detect a minimum clinically significant difference greater than or equal to 8.1 points in the FIQ score. A common standard deviation of 9.6 was assumed, and a rate of loss to follow-up of 0% was estimated, since there were no losses during sample recruitment.
  The chosen standard deviation was that used by Lera (2009)
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2016-01-31 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia impact questionnaire-FIQ | At the begining of the enrolment and 10 weeks later
  FIQ has been validated for the Spanish population. It is a tool for evaluating the impact of FM on physical capacity and quality of life. FIQ scores range: 0 (best functional capacity and quality of life) to 100 (worst state of health). FIQ scores less than 39 are considered to represent a level of slight deterioration, those between 39 and 59 represent moderate deterioration, and scores greater than 59 imply a severe level of disability. The scale comprises 10 items. The first evaluates functional capacity on an ordinal scale from 0(always) to 3(never). The second and third items are numerical scales that evaluate the number of days that participants have been in a good state of health and the number of days in the week on which they have been able to go to do their normal paid work. The other seven items are rated on analogue scales from 0-10 that measure (i)capacity to do a job, (ii)pain, (iii)fatigue, (iv)morning stiffness, (v)muscular numbness, (vi)anxiety and (vii)depression.

SECONDARY OUTCOMES:
Sociodemographic measures | At the begining of the enrolment
  sex, age, civil status, number of children, employment status and level of education. The clinical variables analysed covered the consumption of medication, the number of years that patients had been suffering the symptoms of FMS and the number of years since they had been diagnosed with FMS.

CONTACTS AND LOCATIONS:
Overall Officials: ANNA LLADSER NAVARRO, NR, MsC, Principal Investigator — Institut Investigacio Sanitaria Pere Virgili

IPD SHARING:
Plan to Share IPD: No